CLINICAL TRIAL: NCT03457480
Title: Informing and Correcting Perceptions Regarding Tobacco Products Among Young Adults
Brief Title: Text Messages in Preventing Tobacco Use in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0474; NCI-2018-01277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0474 (Other: M D Anderson Cancer Center); P50CA180906 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (text messages, computer messages) (Experimental): PHASE I: Participants attend focus group over 2 hours.
  PHASE II: Participants receive 2 text messages per day for 30 days at baseline and after 3 months.
  PHASE III: Participants read 64 computer messages with or without images over 30 minutes and have their facial expressions assessed.
  Interventions: Other: Computer-Assisted Intervention; Behavioral: Focus Group; Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Computer-Assisted Intervention — Read computer messages
Behavioral: Focus Group — Attend focus group
Other: Informational Intervention — Receive text messages
Other: Survey Administration — Complete surveys about experience

SUMMARY:
This trial studies how well text messages work in preventing tobacco use in young adults. Text messaging may help to teach young adults about the risks of tobacco products.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess baseline knowledge and risk perceptions about the use of conventional and new and emerging tobacco products among a subset of community college students from the two participating Houston Community College (HCC) campuses (Central and Coleman campuses). (Phase 1.1) II. Test the text messages with university students enrolled in the health communications academic programs. (Phase 1.2) III. Assess the awareness, attitudes, receptivity, and comprehension of the harmful effects of conventional and new and emerging tobacco products among young adults. (Phase 2) IV. Identify the most effective combinations of text message framing for communicating information about the potential harmful effects of tobacco products to young adults. (Phase 2) V. To obtain an objective measure of the psychological (i.e., emotional and cognitive) effect of the messages on young adults. (Phase 3)

EXPLORATORY OBJECTIVES:

I. Define and analyze key moderators of young adult awareness, attitudes, receptivity, and understanding of the harmful risks and constituents of conventional, new and emerging tobacco products. (Phase 2)

OUTLINE:

PHASE I: Participants attend focus group over 2 hours.

PHASE II: Participants receive 2 text messages per day for 30 days at baseline and after 3 months.

PHASE III: Participants read 64 computer messages with or without images over 30 minutes and have their facial expressions assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 (Phase 1, Phase 2, Phase 3)
* Attend classes at either Houston Community College (HCC) Central Campus or Coleman Campus (Phase 1 and Phase 2), Spring Branch Campus (Phase 2) or the University of Houston (Phase 3)
* Own a smartphone capable of receiving texts from the study's text messaging ) resource (Phase 1, Phase 2 and Phase 3)
* Use phone text-messaging features on a regular basis (Phase 1, Phase 2, Phase 3)
* Provide cell phone number (Phase 1, Phase 2, Phase 3)
* Speak and read English (Phase 1, Phase 2, Phase 3)
* Enrolled in a communication program (Phase 1, health communication student review)
* Evidence of smoking susceptibility as defined by the Smoking Susceptibility Scale (Phase 3)

Exclusion Criteria:

-Currently a smoker (Phase 3)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 781 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Baseline knowledge and risk perceptions of Tobacco Use Questionnaire | Up to 8 months
  Participants will take baseline knowledge and risk perceptions about the use of conventional and new and emerging tobacco products among a subset of community college students from the two participating Houston Community College (HCC) campuses (Central and Coleman campuses) Knowledge about whether products contain nicotine scale Yes or No (0-1) A higher score indicates higher knowledge Risk perception for using tobacco products scale from( 1-5) A higher score indicates a higher perception of risk of harm. No scale being used.
Focus Groups Questionnaire | Up to 8 months
  No scale being used. Participants will take part in use of text messages within the university students enrolled in the health communications academic programs. Students will review and rate the messages with the goal of achieving 70% agreement among students across each text message. No scale will be used.
Perceived Risk Perception changes amongst young adults Questionnaire | Up to 8 months
  Participants will show the awareness, attitudes, receptivity, and comprehension of the harmful effects of conventional and new and emerging tobacco products among young adults. 4-point Likert Scale. Higher scores will endorse beliefs for greater benefits of electronic cigarette use. 3-point Likert scale higher score endorse greater addictiveness. Risk perception for using tobacco products. Response format 1-5. A higher score indicates a higher perception of risk of harm. No scale being used.
Information seeking and avoidance about tobacco products Questionnaire | Up to 8 months
  Participants will identify the most effective combinations of text message framing for communicating information about the potential harmful effects of tobacco products to young adults. Risk perception for using tobacco products. Response format 1-5. A Higher score indicates a higher perception of risk of harm. No scale being used.

SECONDARY OUTCOMES:
Risk perceptions related to tobacco products Questionnaire | Up to 8 months
  Participants will have the two-way interactions for synergistic effects on perceived risk for young adults after post 3 month follow up used for determining high and low risk perceptions. Risk perception for using tobacco products. Response format 1-5. A higher score indicates a higher perception of risk of harm. No scale being used.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Prokhorov AV, Calabro KS, Arya A, Russell S, Czerniak KW, Botello GC, Chen M, Yuan Y, Perez A, Vidrine DJ, Perry CL, Khalil GE. Mobile Text Messaging for Tobacco Risk Communication Among Young Adult Community College Students: Randomized Trial of Project Debunk. JMIR Mhealth Uhealth. 2021 Nov 24;9(11):e25618. doi: 10.2196/25618. PMID 34822339
- [Derived] Prokhorov AV, Khalil GE, Calabro KS, Machado TC, Russell S, Czerniak KW, Botello GC, Chen M, Perez A, Vidrine DJ, Perry CL. Mobile Phone Text Messaging for Tobacco Risk Communication Among Young Adult Community College Students: Protocol and Baseline Overview for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 15;7(10):e10977. doi: 10.2196/10977. PMID 30322833
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org